CLINICAL TRIAL: NCT00704912
Title: Treatment of Hyperandrogenism vs. Insulin Resistance in Infertile PCOS Women
Brief Title: Treatment of Hyperandrogenism Versus Insulin Resistance in Infertile Polycystic Ovary Syndrome (PCOS) Women
Acronym: OWL-PCOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Richard S. Legro, M.D., Professor, Obstetrics and Gynecology and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27184
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Orlistat; Contraceptives, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lifestyle intervention (Active Comparator): Orlistat/Meal Replacement/Lifestyle Modification
  Interventions: Drug: Orlistat/Meal Replacement/Lifestyle Modification
- Oral Contraceptives (OCP) (Active Comparator): Loestrin 1/20
  Interventions: Drug: Loestrin 1/20
- Lifestyle/OCP Combined (Active Comparator): Combination of treatments
  Interventions: Drug: Combination of treatments

INTERVENTIONS:
Drug: Orlistat/Meal Replacement/Lifestyle Modification — Orlistat will be given at 60 mg three times per day (1 tablet 3 times a day) before meals, i.e., breakfast, lunch, and dinner.
  Other Names: Orlistat; Alli; Lifestyle Intervention; Weight Loss
  Arms: Lifestyle intervention
Drug: Loestrin 1/20 — Patients will be started on a low dose containing OCP for a continuous 4 month period.
  Other Names: OCP; Oral Contraceptive
  Arms: Oral Contraceptives (OCP)
Drug: Combination of treatments — Medications will be administered as described for the other 2 arms.
  Other Names: Orlistat; Alli; OCP; Oral Contraceptive; Weight Loss; Lifestyle Intervention
  Arms: Lifestyle/OCP Combined

SUMMARY:
The goal of this three-armed randomized controlled trial is to establish the relative roles of treatment of hyperandrogenism versus obesity (as the largest modifiable factor contributing to insulin resistance) in treating infertility and improving pregnancy outcomes among obese PCOS women. The investigators hypothesize that the key to restoring ovulation leading to live birth is to correct hyperandrogenism with oral contraceptive pills, but the key to avoiding later pregnancy complications is to improve insulin sensitivity with weight loss.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is the most common cause of anovulatory infertility among women, and women with PCOS are at increased risk for pregnancy complications such as gestational diabetes and pre-eclampsia. Both hyperandrogenism (HA) and obesity exacerbated insulin resistance (IR) are characteristics of the syndrome, and are targets for treatment, but which should be the predominant focus is still unknown. Phase 1 of this study will be a randomized trial of three preconception interventions in infertile women with PCOS. The first arm will be a combined intervention of medication, meal replacements, and lifestyle modification to improve IR. Orlistat is a gastric lipase inhibitor that reduces the absorption of fat contained in a meal by about 30%. The second arm will be the use of a continuous OCP for 4 months to improve HA. Lo-Estrin 1/20 will be used in a continuous method for 4 months to suppress the ovary. The third arm is the combination of both to improve HA an IR. Phase II of this study will involve ovulation induction with clomiphene citrate with hopeful outcome of pregnancy. Finally, Phase III involve following the pregnancies for outcomes and complications.

ELIGIBILITY:
Couples Inclusion Criteria:

* Partner with sperm concentration of >=14 million/mL in at least one ejaculate with motile sperm.
* Ability to have regular intercourse 2-3 times per week during the ovulation induction phase of study.
* At least one patent tube and normal uterine cavity as determined by sonohysterogram, hysterosalpingogram, or hysteroscopy/laparoscopy within the last 3 years, or confirmation of a intrauterine pregnancy within the past 2 years.
* No previous sterilization procedures(vasectomy, tubal ligation) that have been reversed.
* Wanting to seek pregnancy.

Inclusion Criteria:

* Chronic anovulation or oligomenorrhea defined as intermenstrual periods of >= 45 days or a total of <=8 periods per year.
* Hyperandrogenism will be an elevated total testosterone >=50 ng/dL.
* Hirsutism determined by a modified Ferriman-Gallwey Score >8.
* PCO on ultrasound (12 or more follicles measuring 2-9 mm in diameter).
* BMI >=27 to <=42.
* Normal EKG to rule out any abnormalities with the heart.

Exclusion Criteria:

* Current pregnancy.
* Patients on oral contraceptives, depo progestins, or hormonal implants.
* Patients with hyperprolactinemia defined as two prolactin levels at least one week apart >30 ng/mL.
* Patients with known 21-hydroxylase deficiency by a fasting 17-hydroxyprogesterone (17-OHP) level <2 ng/mL and ACTH stimulation test as needed, or other enzyme deficiency.
* Patients with menopausal FSH levels >20 mIU/mL.
* Patients with uncorrected thyroid disease (TSH <0.45 mIU/ML or >4.5 mIU/ML).
* Patients diagnosed with Type1 or Type II diabetes.
* Patients with liver disease defined as AST or ALT >2 times normal or total bilirubin >2.5 mg/dL.
* Patients with renal disease defined as BUN >30 mg/dL or serum creatinine >1.4 mg/dL.
* Patients with significant anemia (Hemoglobin <10 mg/dL).
* Patients with a history of deep venous thrombosis, pulmonary embolus, or cerebrovascular accident.
* Patients with known heart disease that is likely to be exacerbated by pregnancy.
* Patients with a history of , or suspected cervical carcinoma, endometrial carcinoma, or breast carcinoma. A normal PAP smear or reassuring colposcopy based on current ACOG guidelines will be required.
* Patient with current history of alcohol abuse.
* Patients enrolled simultaneously into other investigative studies.
* Patients taking other medications know to affect reproductive function or metabolism.
* Patients with a suspected adrenal or ovarian tumor secreting androgens.
* Patients with suspected Cushing's syndrome.
* Patients who have undergone a bariatric surgery procedure in the recent past (<12 months).
* Patients with untreated poorly controlled hypertension defined as systolic blood pressure >=150 mm Hg or average diastolic >=100 mm Hg on three measurements obtained 5 minutes apart. If treated, average systolic blood pressure >= 140 mm Hg or average diastolic >= 90 mm Hg.
* Patients with medical conditions that represent contraindications to orlistat, OCP, clomiphene, and/or pregnancy.
* Patients currently participating in lifestyle intervention program (Weight Watchers, Atkins Diet, Curves) or lost more than 5% body weight within the last 6 months.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 217 (Actual)
Dates: Start 2008-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Legro, M.D., Principal Investigator — Penn State College of Medicine, Penn State Milton S. Hershey Medical Center; Christos Coutifaris, M.D., Ph.D., Principal Investigator — Universtiy of Pennsylvania, Department of Obstetrics and Gynecology
Locations (2):
- United States (2):
  - Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Department of Obstetrics and Gynecology, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Steinberg Weiss M, Roe AH, Allison KC, Dodson WC, Kris-Etherton PM, Kunselman AR, Stetter CM, Williams NI, Gnatuk CL, Estes SJ, Sarwer DB, Coutifaris C, Legro RS, Dokras A. Lifestyle modifications alone or combined with hormonal contraceptives improve sexual dysfunction in women with polycystic ovary syndrome. Fertil Steril. 2021 Feb;115(2):474-482. doi: 10.1016/j.fertnstert.2020.08.1396. Epub 2020 Oct 12. PMID 33059886
- [Derived] Shah A, Dodson WC, Kris-Etherton PM, Kunselman AR, Stetter CM, Gnatuk CL, Estes SJ, Allison KC, Sarwer DB, Sluss PM, Coutifaris C, Dokras A, Legro RS. Effects of Oral Contraception and Lifestyle Modification on Incretins and TGF-ss Superfamily Hormones in PCOS. J Clin Endocrinol Metab. 2021 Jan 1;106(1):108-119. doi: 10.1210/clinem/dgaa682. PMID 32968804
- [Derived] Dokras A, Sarwer DB, Allison KC, Milman L, Kris-Etherton PM, Kunselman AR, Stetter CM, Williams NI, Gnatuk CL, Estes SJ, Fleming J, Coutifaris C, Legro RS. Weight Loss and Lowering Androgens Predict Improvements in Health-Related Quality of Life in Women With PCOS. J Clin Endocrinol Metab. 2016 Aug;101(8):2966-74. doi: 10.1210/jc.2016-1896. Epub 2016 Jun 2. PMID 27253669
- [Derived] Legro RS, Dodson WC, Kunselman AR, Stetter CM, Kris-Etherton PM, Williams NI, Gnatuk CL, Estes SJ, Allison KC, Sarwer DB, Diamond MP, Schlaff WD, Casson PR, Christman GM, Barnhart KT, Bates GW, Usadi R, Lucidi S, Baker V, Zhang H, Eisenberg E, Coutifaris C, Dokras A. Benefit of Delayed Fertility Therapy With Preconception Weight Loss Over Immediate Therapy in Obese Women With PCOS. J Clin Endocrinol Metab. 2016 Jul;101(7):2658-66. doi: 10.1210/jc.2016-1659. Epub 2016 May 12. PMID 27172435
- [Derived] Legro RS, Dodson WC, Kris-Etherton PM, Kunselman AR, Stetter CM, Williams NI, Gnatuk CL, Estes SJ, Fleming J, Allison KC, Sarwer DB, Coutifaris C, Dokras A. Randomized Controlled Trial of Preconception Interventions in Infertile Women With Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2015 Nov;100(11):4048-58. doi: 10.1210/jc.2015-2778. Epub 2015 Sep 24. PMID 26401593
- See also: Click here for more information about this study. — http://www.hmc.psu.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 217 subjects consented for the study, of which 149 were randomized to one of the 3 treatment groups. Sixty-eight subjects were not randomized because they withdrew prior to randomization or were determined ineligible during the screening process.
Groups:
- Oral Contraceptives (OCP): Loestrin 1/20: Patients will be started on a low dose containing OCP (20 mcg ethinyl estradiol/1 mg norethindrone acetate daily) for a continuous 4 month period.
Period: Overall Study
Arm/Group | Lifestyle Intervention | Oral Contraceptives (OCP) | Lifestyle/OCP Combined
Started | 50 | 49 | 50
Completed | 44 | 45 | 43
Not Completed | 6 | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle Intervention | Oral Contraceptives (OCP) | Lifestyle/OCP Combined | Total
Number analyzed (Participants) | 50 | 49 | 50 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.6 (3.4) | 29.8 (3.7) | 28.7 (4.2) | 29.0 (3.8)
Gender [Count of Participants; unit: Participants]
  Female | 50 | 49 | 50 | 149
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 5 | 17
  Not Hispanic or Latino | 44 | 43 | 45 | 132
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 7 | 14 | 28
  White | 35 | 40 | 31 | 106
  More than one race | 5 | 2 | 4 | 11
  Unknown or Not Reported | 1 | 0 | 0 | 1
Parity [Number; unit: participants]
  0 births | 41 | 38 | 45 | 124
  >0 births | 9 | 11 | 5 | 25
Weight [Mean (Standard Deviation); unit: kg] | 96.0 (15.8) | 94.6 (14.4) | 95.2 (14.5) | 95.3 (14.8)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 35.1 (4.6) | 35.1 (4.2) | 35.5 (4.4) | 35.2 (4.4)
Metabolic Syndrome [Number; unit: participants]
  Yes | 18 | 14 | 21 | 53
  No | 31 | 34 | 29 | 94
  Unknown | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Live Birth Rate
Time Frame: Participants were followed for 4 months of attempted conception and those who conceived were then followed for the duration of their pregnancy, approximately 9 months.
Measure: Number; unit: participants
Arm/Group | Lifestyle Intervention | Oral Contraceptives (OCP) | Lifestyle/OCP Combined
Number analyzed (Participants) | 50 | 49 | 50
participants | 13 | 5 | 12
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Oral Contraceptives (OCP); Test type: Superiority or Other; p = 0.06, Log-binomial model; Risk Ratio (RR) = 2.5, 95% CI 2-sided [1.0 to 6.6]
Statistical Analysis 2: Comparison: Oral Contraceptives (OCP) vs Lifestyle/OCP Combined; Test type: Superiority or Other; p = 0.08, Log-binomial model; Risk Ratio (RR) = 2.3, 95% CI 2-sided [0.9 to 6.1]
Statistical Analysis 3: Comparison: Lifestyle Intervention vs Lifestyle/OCP Combined; Test type: Superiority or Other; p = 0.82, Log-binomial model; Risk Ratio (RR) = 1.1, 95% CI 2-sided [0.5 to 2.1]

2. Secondary Outcome: Ovulation Rate
Time Frame: Up to 4 months
Measure: Number; unit: total number of ovulations
Units Other Than Participants: Clomiphene Treatment Cycles
Arm/Group | Lifestyle Intervention | Oral Contraceptives (OCP) | Lifestyle/OCP Combined
Number analyzed (Participants) | 50 | 49 | 50
Number analyzed (Clomiphene Treatment Cycles) | 136 | 154 | 140
total number of ovulations | 82 | 71 | 94
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Oral Contraceptives (OCP); Test type: Superiority or Other; p = 0.06, Log-binomial model; Risk Ratio (RR) = 1.3, 95% CI 2-sided [1.0 to 1.7]
Statistical Analysis 2: Comparison: Oral Contraceptives (OCP) vs Lifestyle/OCP Combined; Test type: Superiority or Other; p = 0.002, Log-binomial model; Risk Ratio (RR) = 1.5, 95% CI 2-sided [1.1 to 1.9]
Statistical Analysis 3: Comparison: Lifestyle Intervention vs Lifestyle/OCP Combined; Test type: Superiority or Other; p = 0.28, Log-binomial model; Risk Ratio (RR) = 0.9, 95% CI 2-sided [0.7 to 1.1]

3. Secondary Outcome: Change in Weight
Description: Change from baseline to end of the 4-month intervention.
Time Frame: Baseline, 4 months
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Lifestyle Intervention | Oral Contraceptives (OCP) | Lifestyle/OCP Combined
Number analyzed (Participants) | 50 | 49 | 50
kg | -6.2 [-7.1 to -5.3] | -1.1 [-2.0 to -0.3] | -6.1 [-7.0 to -5.2]
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Oral Contraceptives (OCP); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Difference in Mean Change = -5.0, 95% CI 2-sided [-6.3 to -3.8] — Lifestyle vs. OCP
Statistical Analysis 2: Comparison: Oral Contraceptives (OCP) vs Lifestyle/OCP Combined; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Difference in Mean Change = -5.0, 95% CI 2-sided [-6.2 to -3.7] — Combined vs. OCP
Statistical Analysis 3: Comparison: Lifestyle Intervention vs Lifestyle/OCP Combined; Test type: Superiority or Other; p = 0.92, Mixed Models Analysis; Difference in Mean Change = -0.1, 95% CI 2-sided [-1.3 to 1.2] — Lifestyle vs. Combined

4. Secondary Outcome: Prevalence of Metabolic Syndrome
Time Frame: Baseline, 4 months
Measure: Number; unit: participants
Arm/Group | Lifestyle Intervention | Oral Contraceptives (OCP) | Lifestyle/OCP Combined
Number analyzed (Participants) | 50 | 49 | 50
participants
  Metabolic Syndrome at Baseline | 18 | 14 | 21
  Metabolic Syndrome at End of Intervention | 18 | 21 | 16
Statistical Analysis 1: Comparison: Lifestyle Intervention; Comparing change in prevalence of metabolic syndrome from baseline to the end of intervention; Test type: Superiority or Other; p = 0.60, GEE; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.6 to 2.2] — End of intervention compared to baseline
Statistical Analysis 2: Comparison: Oral Contraceptives (OCP); Comparing change in prevalence of metabolic syndrome from baseline to the end of intervention; Test type: Superiority or Other; p = 0.001, GEE; Odds Ratio (OR) = 2.5, 95% CI 2-sided [1.4 to 4.3] — End of intervention compared to baseline
Statistical Analysis 3: Comparison: Lifestyle/OCP Combined; Comparing change in prevalence of metabolic syndrome from baseline to the end of intervention; Test type: Superiority or Other; p = 0.18, GEE; Odds Ratio (OR) = 0.7, 95% CI 2-sided [0.4 to 1.2] — End of intervention compared to baseline
Statistical Analysis 4: Comparison: Lifestyle Intervention vs Oral Contraceptives (OCP); Test type: Superiority or Other; p = 0.08, GEE
Statistical Analysis 5: Comparison: Oral Contraceptives (OCP) vs Lifestyle/OCP Combined; Test type: Superiority or Other; p = 0.001, GEE
Statistical Analysis 6: Comparison: Lifestyle Intervention vs Lifestyle/OCP Combined; Test type: Superiority or Other; p = 0.22, GEE

ADVERSE EVENTS:
Arm/Group | Lifestyle Intervention | Oral Contraceptives (OCP) | Lifestyle/OCP Combined
Serious Adverse Events (participants affected / at risk) | 3/50 | 0/49 | 1/50
Other Adverse Events (participants affected / at risk) | 32/50 | 37/49 | 43/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lifestyle Intervention (N=50) | Oral Contraceptives (OCP) (N=49) | Lifestyle/OCP Combined (N=50)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) — Episode of abnormal uterine bleeding leading to ER visit
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) — Ectopic pregnancy requiring surgery
Preterm delivery (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) — Preterm delivery of twins at 20 weeks: 1 live birth and 1 IUFD secondary to infection
Perforated appendix (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Postpartum hospitalization for perforated appendix
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Lifestyle Intervention (N=50) | Oral Contraceptives (OCP) (N=49) | Lifestyle/OCP Combined (N=50)
Steatorrhea/Diarrhea (Gastrointestinal disorders) | 6 | 0 | 12 — Phase I Intervention
Headache (General disorders) | 15 | 14 | 18 — Phase I Intervention
Upper Respiratory Infections (Respiratory, thoracic and mediastinal disorders) | 8 | 8 | 13 — Phase I Intervention
Nausea/Vomiting (General disorders) | 6 | 7 | 9 — Phase I Intervention
Breast Pain (Reproductive system and breast disorders) | 1 | 10 | 6 — Phase I Intervention
Abdominal Pain (General disorders) | 5 | 1 | 10 — Phase I Intervention
Dysmenorrhea (Reproductive system and breast disorders) | 1 | 8 | 3 — Phase I Intervention
Constipation (Gastrointestinal disorders) | 6 | 1 | 4 — Phase I Intervention
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 | 4 | 6 — Phase I Intervention
Mood Swings (Psychiatric disorders) | 3 | 3 | 3 — Phase I Intervention
Gas/Bloating (Gastrointestinal disorders) | 2 | 2 | 5 — Phase I Intervention
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 4 — Phase I Intervention
Vaginitis/Vulvitis (Reproductive system and breast disorders) | 1 | 4 | 1 — Phase I Intervention
Pelvic Pain (Reproductive system and breast disorders) | 2 | 3 | 1 — Phase I Intervention
Dry Mouth (General disorders) | 4 | 0 | 1 — Phase I Intervention
Dizziness/Vertigo (General disorders) | 3 | 2 | 0 — Phase I Intervention
Fatigue (General disorders) | 1 | 2 | 3 — Phase I Intervention
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 — Phase I Intervention
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 3 — Phase I Intervention
Insomnia (General disorders) | 2 | 0 | 3 — Phase I Intervention
Tachycardia (General disorders) | 1 | 0 | 3 — Phase I Intervention
Pelvic Pain (Reproductive system and breast disorders) | 7/44 | 12/44 | 13/43 — Phase II Ovulation Induction
Headache (General disorders) | 4/44 | 6/44 | 12/43 — Phase II Ovulation Induction
Breast Pain (Reproductive system and breast disorders) | 5/44 | 7/44 | 9/43 — Phase II Ovulation Induction
Hot flushes (Reproductive system and breast disorders) | 4/44 | 6/44 | 3/43 — Phase II Ovulation Induction
Nausea/Vomiting (General disorders) | 5/44 | 3/44 | 5/43 — Phase II Ovulation Induction
Upper Respiratory Infections (Respiratory, thoracic and mediastinal disorders) | 2/44 | 5/44 | 5/43 — Phase II Ovulation Induction
Mood Swings (Psychiatric disorders) | 3/44 | 3/44 | 2/43 — Phase II Ovulation Induction
Dysmenorrhea (Reproductive system and breast disorders) | 1/44 | 6/44 | 1/43 — Phase II Ovulation Induction
Gas/Bloating (Gastrointestinal disorders) | 4/44 | 1/44 | 3/43 — Phase II Ovulation Induction
Constipation (Gastrointestinal disorders) | 2/44 | 2/44 | 3/43 — Phase II Ovulation Induction
Fatigue (General disorders) | 2/44 | 1/44 | 3/43 — Phase II Ovulation Induction
Abdominal Pain (General disorders) | 2/44 | 3/44 | 1/43 — Phase II Ovulation Induction
Visual Changes (General disorders) | 1/44 | 0/44 | 3/43 — Phase II Ovulation Induction
Vaginal Dryness/Pain (Reproductive system and breast disorders) | 0/44 | 3/44 | 0/43 — Phase II Ovulation Induction
Nausea/Vomiting (Pregnancy, puerperium and perinatal conditions) | 4/16 | 0/8 | 1/14 — Phase III After Conception: First trimester
Fatigue (Pregnancy, puerperium and perinatal conditions) | 3/16 | 0/8 | 1/14 — Phase III After Conception: First trimester
Pelvic Pain (Pregnancy, puerperium and perinatal conditions) | 3/16 | 0/8 | 1/14 — Phase III After Conception: First trimester
Breast Pain (Pregnancy, puerperium and perinatal conditions) | 1/16 | 0/8 | 2/14 — Phase III After Conception: First trimester
Headache (Pregnancy, puerperium and perinatal conditions) | 2/16 | 0/8 | 1/14 — Phase III After Conception: First trimester
Mood Swings (Pregnancy, puerperium and perinatal conditions) | 1/16 | 0/8 | 1/14 — Phase III After Conception: First trimester
Constipation (Pregnancy, puerperium and perinatal conditions) | 1/16 | 0/8 | 1/14 — Phase III After Conception: First trimester
Hot flushes (Pregnancy, puerperium and perinatal conditions) | 2/16 | 0/8 | 0/14 — Phase III After Conception: First trimester
Spotting in pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/16 | 0/8 | 1/14 — Phase III After Conception: First trimester
Hypertension (Pregnancy, puerperium and perinatal conditions) | 1/16 | 0/8 | 0/14 — Phase III After Conception: First trimester
Vaginitis/Vulvitis (Pregnancy, puerperium and perinatal conditions) | 1/16 | 0/8 | 0/14 — Phase III After Conception: First trimester
Vaginal Dryness/Pain (Pregnancy, puerperium and perinatal conditions) | 1/16 | 0/8 | 0/14 — Phase III After Conception: First trimester
Hyperemesis (Pregnancy, puerperium and perinatal conditions) | 1/16 | 0/8 | 0/14 — Phase III After Conception: First trimester
Urinary tract infection in pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/16 | 0/8 | 0/14 — Phase III After Conception: First trimester
Dizziness/Vertigo (Pregnancy, puerperium and perinatal conditions) | 0/16 | 0/8 | 1/14 — Phase III After Conception: First trimester
Rash (Pregnancy, puerperium and perinatal conditions) | 0/16 | 1/8 | 0/14 — Phase III After Conception: First trimester
Gas/Bloating (Pregnancy, puerperium and perinatal conditions) | 1/16 | 0/8 | 0/14 — Phase III After Conception: First trimester
Abdominal Pain (Pregnancy, puerperium and perinatal conditions) | 1/16 | 0/8 | 0/14 — Phase III After Conception: First trimester
Dyspepsia (Pregnancy, puerperium and perinatal conditions) | 0/16 | 0/8 | 1/14 — Phase III After Conception: First trimester
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 4/16 | 1/8 | 2/14 — Phase III After Conception: Second and Third trimester
Gestational Diabetes (Pregnancy, puerperium and perinatal conditions) | 3/16 | 1/8 | 2/14 — Phase III After Conception: Second and Third trimester
Preterm Delivery (Pregnancy, puerperium and perinatal conditions) | 3/16 | 0/8 | 0/14 — Phase III After Conception: Second and Third trimester
Premature Rupture of Membranes (Pregnancy, puerperium and perinatal conditions) | 3/16 | 0/8 | 0/14 — Phase III After Conception: Second and Third trimester
Upper Respiratory Infections (Pregnancy, puerperium and perinatal conditions) | 3/16 | 0/8 | 0/14 — Phase III After Conception: Second and Third trimester
Placental Abnormalities (Pregnancy, puerperium and perinatal conditions) | 1/16 | 1/8 | 0/14 — Phase III After Conception: Second and Third trimester
Dental abscess (Pregnancy, puerperium and perinatal conditions) | 1/16 | 0/8 | 0/14 — Phase III After Conception: Second and Third trimester
Dental, other (Pregnancy, puerperium and perinatal conditions) | 1/16 | 0/8 | 0/14 — Phase III After Conception: Second and Third trimester
Other specified disorders of biliary tract (Pregnancy, puerperium and perinatal conditions) | 0/16 | 0/8 | 1/14 — Phase III After Conception: Second and Third trimester
Breast lump (Pregnancy, puerperium and perinatal conditions) | 0/16 | 0/8 | 1/14 — Phase III After Conception: Second and Third trimester
Vaginitis/Vulvitis (Pregnancy, puerperium and perinatal conditions) | 0/16 | 0/8 | 1/14 — Phase III After Conception: Second and Third trimester
Urinary tract infection in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/16 | 0/8 | 1/14 — Phase III After Conception: Second and Third trimester
Incompetent cervix (Pregnancy, puerperium and perinatal conditions) | 1/16 | 0/8 | 0/14 — Phase III After Conception: Second and Third trimester
Infection of amniotic cavity (Pregnancy, puerperium and perinatal conditions) | 0/16 | 0/8 | 1/14 — Phase III After Conception: Second and Third trimester
Pruritus (Pregnancy, puerperium and perinatal conditions) | 0/16 | 0/8 | 1/14 — Phase III After Conception: Second and Third trimester
Dizziness/Vertigo (Pregnancy, puerperium and perinatal conditions) | 0/16 | 1/8 | 0/14 — Phase III After Conception: Second and Third trimester
Sleep disturbance (Pregnancy, puerperium and perinatal conditions) | 1/16 | 0/8 | 0/14 — Phase III After Conception: Second and Third trimester
Sleep apnea (Pregnancy, puerperium and perinatal conditions) | 1/16 | 0/8 | 0/14 — Phase III After Conception: Second and Third trimester
Edema localized (Pregnancy, puerperium and perinatal conditions) | 1/16 | 0/8 | 0/14 — Phase III After Conception: Second and Third trimester
Glycosuria (Pregnancy, puerperium and perinatal conditions) | 1/16 | 0/8 | 0/14 — Phase III After Conception: Second and Third trimester
Headache (Pregnancy, puerperium and perinatal conditions) | 0/16 | 0/8 | 1/14 — Phase III After Conception: Second and Third trimester
Musculoskeletal Pain (Pregnancy, puerperium and perinatal conditions) | 0/16 | 0/8 | 1/14 — Phase III After Conception: Second and Third trimester
Pregnancy-induced Hypertension (Pregnancy, puerperium and perinatal conditions) | 2/16 | 0/8 | 0/14 — Delivery and Postpartum
Pulmonary collapse (Pregnancy, puerperium and perinatal conditions) | 1/16 | 0/8 | 0/14 — Delivery and Postpartum
Postpartum depression (Pregnancy, puerperium and perinatal conditions) | 0/16 | 1/8 | 0/14 — Delivery and Postpartum
Postpartum infection (Pregnancy, puerperium and perinatal conditions) | 1/16 | 0/8 | 0/14 — Delivery and Postpartum
Neonatal Jaundice (Pregnancy, puerperium and perinatal conditions) | 2/12 | 1/5 | 4/12 — After 20 weeks pregnancy in fetus through neonatal period
Intrauterine growth restriction (Pregnancy, puerperium and perinatal conditions) | 1/12 | 0/5 | 1/12 — After 20 weeks pregnancy in fetus through neonatal period
Neonatal infection (Pregnancy, puerperium and perinatal conditions) | 0/12 | 0/5 | 1/12 — After 20 weeks pregnancy in fetus through neonatal period
Other complication of infant after delivery (Pregnancy, puerperium and perinatal conditions) | 0/12 | 0/5 | 1/12 — After 20 weeks pregnancy in fetus through neonatal period

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No